CLINICAL TRIAL: NCT05219487
Title: Investigating NMJ Defects in SMA Following Central and Peripheral SMN Restoration
Status: Recruiting | Type: Observational
Sponsor: Bakri Elsheikh (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Bakri Elsheikh, Professor of Neurology, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2021H0158; ML43109 (Other: Genentech, Inc.)
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Risdiplam — Risdiplam is administered orally once daily and the recommended dosage is determined by age and body weight (see Table 1) [as outlined in the US Prescribing Information for EVRYSDI™(risdiplam)].
  Table 1 Adult and Pediatric Dosing Regimen by Age and Body Weight: US Prescribing Information
  Age and Body Weight (Recommended Daily Dosage): 2 months to less than 2 years of age (0.2 mg/kg); 2 years of age and older weighing less than 20 kg (0.25 mg/kg); 2 years of age and older weighing 20 kg or more (5 mg)
  Other Names: Evrysdi®

SUMMARY:
This is an observational study to investigate the improvement of NMJ defects in adult patients with SMA following treatment with Risdiplam. Eligible patients will have received treatment with daily oral Risdiplam after receiving approval through their commercial insurance or drug assistance program. All subjects will be evaluated at one visit. Eligible subjects must have been receiving risdiplam for at least 12 months.

DETAILED DESCRIPTION:
This is a proof of concept trial to investigate the impact of FDA approved therapy for adults with SMA on NMJ transmission. The study will enroll genetically confirmed adults with 5 q SMA treated with risdiplam for at least 12 months. Dosing will be weight- based as approved by the FDA (US Prescribing Information).

Assessments will include medical history, general physical and neurological examinations, vital signs, and the recording of adverse events. Diagnostic tests will include repetitive nerve stimulation (RNS), motor unit number estimation (MUNE), and decomposition EMG (dEMG). Further evaluations will utilize the Hammersmith Functional Motor Scale Expanded (HFMSE), the Revised Upper Limb Module (RULM), the modified SMA Functional Rating Scale (SMAFRS), and the Fatigue Severity Scale (FSS). For ambulatory subjects, the assessment will include a six-minute walk test, while for non-ambulatory subjects, the Children's Hospital of Philadelphia Adult/Adolescent Test of Neuromuscular Disorders (CHOP INTEND) will be performed. Handheld dynamometry will be used to measure strength in bilateral shoulder abduction, elbow flexion, elbow extension, hip flexion, hip abduction, hip adduction, knee flexion, and knee extension.

The study aims to investigate the impact of Risdiplam on neuromuscular junction (NMJ) function by assessing changes in the percent decrement of the compound muscle action potential amplitude, as measured through 3 Hz repetitive nerve stimulation (RNS) of the spinal accessory nerve. These results will be compared to historical controls. Additionally, the study will evaluate the differences in strength, motor function, and electrophysiological test scores between groups, which will be stratified based on a 10% decrement cutoff. Further analysis will explore the association between these measures and percent decrement among ambulatory and non-ambulatory patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age 18-70 years at time of signing Informed Consent Form
* Able and willing to provide written informed consent and to comply with the program protocol according to ICH and local regulations
* Ability to comply with the study protocol, in the investigator's judgment
* Adequately recovered from any acute illness at the time of screening, and considered clinically well enough to participate, in the opinion of the treating physician
* Patients with retinopathy of prematurity should have evidence of stable disease
* Genetic confirmation of 5q SMA documented on standard genetic tests for the disorder
* Treated with risdiplam for a duration of 12 months or longer

Exclusion Criteria:

* Treatment with an investigational therapy within 180 days prior to initiation of study drug
* History of established diagnosis of neuromuscular junction disorder
* Co-morbid conditions that preclude travel or testing
* Patients who are, in the investigator's opinion, mentally or legally incapacitated to provide an informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll genetically confirmed adults with 5 q SMA with electrodiagnostic evidence of NMJ defects treated with risdiplam for a duration of 12 months or longer.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Decrement on repetitive nerve stimulation | Baseline
  Change in the percent decrement of the compound muscle action potential amplitude assessed using 3 Hz repetitive nerve stimulation (RNS) of the spinal accessory nerve compared to historical controls.
  If CMAP amplitude is absent at spinal accessory nerve, SMA, ulnar CMAP will be used to assess NMJ transmission.

SECONDARY OUTCOMES:
Six Minute Walk Test (6MWT) Total Distance | Baseline
  The score difference between groups stratified using a 10% decrement cutoff
Six Minute Walk Test Difference in Distance Between the First and Final minute | Baseline
  The score difference between groups stratified using a 10% decrement cutoff
Modified Spinal Muscular Atrophy Function Rating Scale (SMA-FRS) | Baseline
  The score difference between groups stratified using a 10% decrement cutoff (scale 0-40, higher score is better).
Revised Upper Limb Module (RULM) | Baseline
  The score difference between groups stratified using a 10% decrement cutoff (scale 0-37, a higher score is better)
Hammersmith Functional Rating Scale (HFMSE) | Baseline
  The score difference between groups stratified using a 10% decrement cutoff (0-66, a higher score is better
Fatigue Severity Scale (FSS) | Baseline
  The score difference between groups stratified using a 10% decrement cutoff (9-63, the higher the score the higher the fatigue)
Children's Hospital of Philadelphia - Adult Test of Neuromuscular Disorders (CHOP-ATEND) | Baseline
  The score difference between groups stratified using a 10% decrement cutoff analyses (0-52, a higher score is better)
Strength Measure using Hand Held Dynamometry | Baseline
  Strength measurements of of bilateral shoulder abduction, elbow flexion, elbow extension, hip flexion, hip abduction, hip adduction, knee flexion and knee extension. The score difference between groups stratified using a 10% decrement cutoff analyses.
Ulnar Compound Muscle Action Potential (Ulnar -CMAP) | Baseline
  The difference in amplitudes between groups stratified using a 10% decrement cutoff
Motor Unit Number Estimation (MUNE) | Baseline
  Ulnar MUNE using modified multipoint technique. The difference in MUNE score between groups stratified using a 10% decrement cutoff

CONTACTS AND LOCATIONS:
Overall Officials: Bakri Elsheikh, MBBS, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States